CLINICAL TRIAL: NCT05782946
Title: The Effect of Heavy Smoking on Early Post Operative Cognitive Dysfunction in Senile Patients After Urological Day-case Surgery , A Randomized Controlled Trial .
Brief Title: The Effect of Heavy Smoking on Early Post Operative Cognitive Dysfunction in Senile Patients .
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahmoud Hussein Bahr, Associated Professor of Anesthesiology and Surgical Intensive Care and pain medicine, Beni-Suef University
Other Study IDs: FMBSUREC/12022023/Emam
Record Dates: First submitted 2023-02-15; First posted 2023-03-24 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Smoking and POCD
Keywords: Postoperative Cognitive Dysfunction; Smoking; General Anaesthesia; Day-case surgery
MeSH Terms: conditions — Smoking; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cognitive dysfunction is the impairment of mental process of perception, memory and information processing which allow the human to acquire knowledge and plan for the future . The etiology of Postoperative cognitive dysfunction (POCD) is unclear and seems to be multifactorial involving a combination of patient, surgical, anesthetic and environmental factors .It can be a manifestation of transient or permanent cerebral injury. While cognitive function tends to improve over months to years postoperatively in affected individuals, some proportion has seemingly permanent cognitive injury .

DETAILED DESCRIPTION:
Cognitive dysfunction is the impairment of mental process of perception, memory and information processing which allow the human to acquire knowledge and plan for the future . The etiology of Postoperative cognitive dysfunction (POCD) is unclear and seems to be multifactorial involving a combination of patient, surgical, anesthetic and environmental factors .It can be a manifestation of transient or permanent cerebral injury. While cognitive function tends to improve over months to years postoperatively in affected individuals, some proportion has seemingly permanent cognitive injury .

Most of the studies of POCD, however, have methodological difficulties, as pointed out by Newman and colleagues in their review of more than 40 studies . a major difficulty in trying to compare investigations or establish an incidence of POCD was the diversity in participants, types of surgery and anesthesia, methods of assessment, definition of POCD, and mode of analysis .

The number of tobacco smokers has been decreasing over the last decade in most Western countries, while the percentage of smokers is still increasing in some developing countries . Tobacco smoking is still one of the major causes of mortality and morbidity worldwide . In particular, it is well known that smoking is strongly associated with cardiovascular diseases, pulmonary diseases and cancer. In addition, it is also thought that smoking could increase the risk of poor postoperative outcomes, in ways including impaired wound healing ، infections and cardiopulmonary complications.

The definition of day surgery in Great Britain and Ireland is clear; the patient is admitted and discharged on the same day, with day surgery as the intended management. The term '23-h stay' is used in the United states healthcare system .

ELIGIBILITY:
Inclusion Criteria:

* patients between 65 & 80 ys
* elective urological day-case surgery
* ASA physical status 1

Exclusion Criteria:

* Patients not ASA1
* Patients receiving sedatives as midazolam.
* Pregnant Patients .
* Patients with cerebrovascular diseases .
* Patients with history of drug allergy or patients with substance abuse .
* Time of anesthesia less than 30 minute ,or more than one hour .
* Irrigation fluid rather than warm saline(40 degree ) or volume more than 1500 ml
* post- secondary Education level .

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Senile patients 65 : 80 ys Chronic heavy smokers & non smokers ASA physical status 1
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | MoCA was performed preoperative .
  Montreal Cognitive Assessment (MoCA) MoCA was a questionaire performed preoperative then post operative . The MoCA used in this study was developed by Professor Nasreddine in 2004 and is used for the rapid screening assessment of mild cognitive impairment. The cognitive areas assessed by MoCA included attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, calculation and orientation. The scale had a total score of 30 points. ≥26 points were considered as having no cognitive impairment .
Montreal Cognitive Assessment (MoCA) | 1 hour Postoperative
  Montreal Cognitive Assessment (MoCA) MoCA was a questionnaire performed preoperative then post operative . The MoCA used in this study was developed by Professor Nasreddine in 2004 and is used for the rapid screening assessment of mild cognitive impairment. The cognitive areas assessed by MoCA included attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, calculation and orientation. The scale had a total score of 30 points. ≥26 points were considered as having no cognitive impairment .
Montreal Cognitive Assessment (MoCA) | 6 hours post operative .
  Montreal Cognitive Assessment (MoCA) MoCA was a questionnaire performed preoperative then post operative. The MoCA used in this study was developed by Professor Nasreddine in 2004 and is used for the rapid screening assessment of mild cognitive impairment. The cognitive areas assessed by MoCA included attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, calculation and orientation. The scale had a total score of 30 points. ≥26 points were considered as having no cognitive impairment .
Montreal Cognitive Assessment (MoCA) | 24 hours post operative.
  Montreal Cognitive Assessment (MoCA) MoCA was a questionnaire performed preoperative then post operative . The MoCA used in this study was developed by Professor Nasreddine in 2004 and is used for the rapid screening assessment of mild cognitive impairment. The cognitive areas assessed by MoCA included attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, calculation and orientation. The scale had a total score of 30 points. ≥26 points were considered as having no cognitive impairment .

SECONDARY OUTCOMES:
age , in years . | Preoperatively
  age , in years .
heart rate ( beat / minute ) | Preoperatively and every 15 minutes for 3 hours .
  heart rate ( beat / minute )
Body mass index( BMI ) = weight in kg/ height in m^2 . | Preoperatively.
  Body mass index( BMI ) = weight in kg/ height in m^2 .
Mean arterial blood pressure ,MAP, ( mmHg ) | Preoperatively and every 15 minutes for 3 hours .
  Mean arterial blood pressure ,MAP, ( mmHg )
peripheral oxygen saturation (Spo2) | Preoperatively and every 15 minutes for 3 hours .
  peripheral oxygen saturation (Spo2)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud H Bahr, Principal Investigator — Faculty of Medicine Beni-Suef University Egypt
Locations (1):
- Faculty of medicine.Beni-suef university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet